CLINICAL TRIAL: NCT02777749
Title: Adductor Canal Block Versus Periarticular Bupivicaine Injection in Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Jeffrey Geller, Associate Professor of Orthopedic Surgery at the Columbia University Medical Center, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AAAQ0850
Record Dates: First submitted 2016-05-11; First posted 2016-05-19 (Estimated); Results first posted 2019-03-20 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Adductor Canal Block (Active Comparator): 15 cc's of 0.5% bupivacaine preoperatively administered by the regional pain anesthesia team in the pre-operative block area, just prior to surgery.
  Adductor Canal Block (ACB)
  Interventions: Drug: Bupivacaine
- Periarticular SB (Active Comparator): 50 cc's of 0.25% bupivacaine will be injected intraoperatively, just prior to wound closure, by the performing surgeon.
  Interventions: Drug: Bupivacaine
- ACB + SB (Active Comparator): 15 cc's of 0.5% bupivacaine preoperatively administered by the regional pain anesthesia team in the pre-operative block area, just prior to surgery.
  50 cc's of 0.25% bupivacaine will be injected intraoperatively, just prior to wound closure, by the performing surgeon.
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Bupivacaine — 15 cc's of 0.5% bupivacaine or 50 cc's of 0.25% short-acting bupivacaine (SB), intramuscular injection
  Other Names: Bupivacaine Hydrochloride; Marcaine

SUMMARY:
The objective of the study is to compare the efficacy of adductor canal blocks versus periarticular bupivacaine injections for pain management in total knee arthroplasty. This randomized clinical trial will compare outcomes between adductor canal blocks, periarticular bupivacaine injections, and periarticular liposomal bupivacaine injections. Results from this study will help determine the most appropriate perioperative pain management strategy for patients undergoing a total knee arthroplasty.

DETAILED DESCRIPTION:
Over 600,000 total knee arthroplasties (TKAs) are performed each year in the United States, with expectations for greater than 4 million/year by the year 2030. Since the onset of TKAs in the 1960's, there have been developments that have improved both functionality and patient satisfaction. In the last decade, a focus has been made on multimodal pain management protocols, more rapid functional recovery, reduced length of hospital stay, and minimizing side effects of treatment while maintaining function and durability. The widespread use of regional anesthesia has led to improvements in pain control, more rapid functional recovery, and reduced length of stay. In recent years many surgeons have transitioned from femoral nerve blocks (proximal femoral nerve) to adductor canal blocks (distal femoral nerve) to maintain a sensory block for pain control, while minimizing any motor blockade that is typically seen in proximal femoral nerve blocks, which would hamper rehabilitation, and increase risk of falls. In addition to regional blocks, which are typically performed in the preoperative setting, some surgeons favor an intraoperative periarticular anesthetic injection (PAI), typically with bupivacaine or the long acting form liposomal bupivacaine, either in conjunction with an adductor canal block, or independently. In theory, PAI has the advantage of a comparable sensory nerve block as an adductor canal block, without the disadvantages and risks, which include prolonged quadriceps weakness, fall risk, and neurologic dysfunction.

The purpose of this randomized control trial is to compare the efficacy of adductor canal blocks versus periarticular bupivacaine injections for pain management in total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

- Patients undergoing an unilateral primary total knee arthroplasty under the care of the two senior arthroplasty surgeons.

Exclusion Criteria:

- Allergy to bupivicaine or liposomal bupivicaine.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2016-07-19 (Actual); Primary Completion 2017-09-19 (Actual); Study Completion 2017-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Geller, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cram P, Lu X, Kates SL, Singh JA, Li Y, Wolf BR. Total knee arthroplasty volume, utilization, and outcomes among Medicare beneficiaries, 1991-2010. JAMA. 2012 Sep 26;308(12):1227-36. doi: 10.1001/2012.jama.11153. PMID 23011713
- [Background] Berend ME, Berend KR, Lombardi AV Jr. Advances in pain management: game changers in knee arthroplasty. Bone Joint J. 2014 Nov;96-B(11 Supple A):7-9. doi: 10.1302/0301-620X.96B11.34514. PMID 25381400
- [Background] Paul JE, Arya A, Hurlburt L, Cheng J, Thabane L, Tidy A, Murthy Y. Femoral nerve block improves analgesia outcomes after total knee arthroplasty: a meta-analysis of randomized controlled trials. Anesthesiology. 2010 Nov;113(5):1144-62. doi: 10.1097/ALN.0b013e3181f4b18. PMID 20966667
- [Background] Grevstad U, Mathiesen O, Valentiner LS, Jaeger P, Hilsted KL, Dahl JB. Effect of adductor canal block versus femoral nerve block on quadriceps strength, mobilization, and pain after total knee arthroplasty: a randomized, blinded study. Reg Anesth Pain Med. 2015 Jan-Feb;40(1):3-10. doi: 10.1097/AAP.0000000000000169. PMID 25376972
- [Background] Wang C, Cai XZ, Yan SG. Comparison of Periarticular Multimodal Drug Injection and Femoral Nerve Block for Postoperative Pain Management in Total Knee Arthroplasty: A Systematic Review and Meta-Analysis. J Arthroplasty. 2015 Jul;30(7):1281-6. doi: 10.1016/j.arth.2015.02.005. Epub 2015 Feb 20. PMID 25735501
- [Background] Schroer WC, Diesfeld PG, LeMarr AR, Morton DJ, Reedy ME. Does Extended-Release Liposomal Bupivacaine Better Control Pain Than Bupivacaine After Total Knee Arthroplasty (TKA)? A Prospective, Randomized Clinical Trial. J Arthroplasty. 2015 Sep;30(9 Suppl):64-7. doi: 10.1016/j.arth.2015.01.059. Epub 2015 Jun 3. PMID 26117072
- [Background] Berry J. Audience response-practice norm/trends. 22nd Annual Meeting of the American Association of Hip and Knee Surgeons. American Association of Hip and Knee Surgeons. November 2012.

RESULTS

PARTICIPANT FLOW:
Groups:
- Adductor Canal Block: 15 cc's of 0.5% bupivacaine preoperatively administered by the regional pain anesthesia team in the pre-operative block area, just prior to surgery.
  Adductor Canal Block (ACB)
  Bupivacaine: 15 cc's of 0.5% bupivacaine or 20 cc's short-acting bupivacaine (SB), intramuscular injection
- Periarticular SB: 50 cc's of bupivacaine will be injected intraoperatively, just prior to wound closure, by the performing surgeon.
  Bupivacaine: 15 cc's of 0.5% bupivacaine or 50 cc's short-acting bupivacaine (SB), intramuscular injection
- ACB + SB: 15 cc's of 0.5% bupivacaine preoperatively administered by the regional pain anesthesia team in the pre-operative block area, just prior to surgery.
  50 cc's of bupivacaine will be injected intraoperatively, just prior to wound closure, by the performing surgeon.
  Bupivacaine: 15 cc's of 0.5% bupivacaine or 50 cc's short-acting bupivacaine (SB), intramuscular injection
Period: Overall Study
Arm/Group | Adductor Canal Block | Periarticular SB | ACB + SB
Started | 53 | 51 | 51
Completed | 53 | 51 | 51
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Periarticular SB: 20 cc's of bupivacaine will be injected intraoperatively, just prior to wound closure, by the performing surgeon.
  Bupivacaine: 15 cc's of 0.5% bupivacaine or 20 cc's short-acting bupivacaine (SB), intramuscular injection
- ACB + SB: 15 cc's of 0.5% bupivacaine preoperatively administered by the regional pain anesthesia team in the pre-operative block area, just prior to surgery.
  20 cc's of bupivacaine will be injected intraoperatively, just prior to wound closure, by the performing surgeon.
  Bupivacaine: 15 cc's of 0.5% bupivacaine or 20 cc's short-acting bupivacaine (SB), intramuscular injection
- Total: Total of all reporting groups
Arm/Group | Adductor Canal Block | Periarticular SB | ACB + SB | Total
Number analyzed (Participants) | 53 | 51 | 51 | 155
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 9 | 13 | 36
  >=65 years | 39 | 42 | 38 | 119
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (10) | 73 (10) | 71 (10) | 71 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 33 | 37 | 108
  Male | 15 | 18 | 14 | 47
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change in VAS Pain Scores
Description: Post-operatively, visual analog scale (VAS) pain scores will be recorded two times/day from Post-Operative Day (POD) 0 through POD3. VAS Scores range from 0 to 10, with 0 being "No Pain" and 10 being the "Worst Pain"
Time Frame: Day 0 through Day 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- ACB + SB: 15 cc's of 0.5% bupivacaine preoperatively administered by the regional pain anesthesia team in the pre-operative block area, just prior to surgery.
  50 cc's of bupivacaine will be injected intraoperatively, just prior to wound closure, by the performing surgeon.
  Bupivacaine: 15 cc's of 0.5% bupivacaine or 20 cc's short-acting bupivacaine (SB), intramuscular injection
Arm/Group | Adductor Canal Block | Periarticular SB | ACB + SB
Number analyzed (Participants) | 53 | 51 | 51
scores on a scale
  Day 0 | 3.0 (2.9) | 3.0 (3.0) | 2.7 (2.6)
  Day 1 | 3.9 (2.3) | 3.8 (2.4) | 3.0 (2.1)
  Day 2 | 4.1 (2.5) | 3.8 (2.4) | 3.3 (2.5)
  Day 3 | 4.2 (3.1) | 3.0 (2.8) | 2.0 (2.0)

2. Secondary Outcome: Change in Activity Level
Description: Daily steps taken will be recorded. The more steps taken daily the better. Minimum is 0 steps, maximum is unlimited.
Time Frame: Day 0 and Day 1
Measure: Mean (Standard Deviation); unit: steps
Groups:
- Periarticular SB: 50 cc's of bupivacaine will be injected intraoperatively, just prior to wound closure, by the performing surgeon.
  Bupivacaine: 15 cc's of 0.5% bupivacaine or 20 cc's short-acting bupivacaine (SB), intramuscular injection
Arm/Group | Adductor Canal Block | Periarticular SB | ACB + SB
Number analyzed (Participants) | 53 | 51 | 51
steps
  Day 0 | 26 (33) | 68 (63) | 65 (50)
  Day 1 | 124 (117) | 120 (117) | 139 (118)

3. Secondary Outcome: Opioid Consumption
Description: Total amount of opioid consumption post-operatively will be recorded. The less opioids consumed (mg) postoperatively the better. A morphine equivalence metric will be used for equianalgesic comparison. Minimum is 0 mg, maximum is unlimited.
Time Frame: Day 0 through Day 3
Measure: Mean (Standard Deviation); unit: morphine equivalents
Arm/Group | Adductor Canal Block | Periarticular SB | ACB + SB
Number analyzed (Participants) | 53 | 51 | 51
morphine equivalents
  Combined (POD0 through POD3) | 131 (74) | 100 (62) | 98 (62)
  POD0 | 33 (15) | 31 (18) | 35 (21)
  POD1 | 48 (25) | 42 (31) | 40 (30)
  POD2 | 35 (29) | 20 (22) | 18 (21)
  POD3 | 13 (23) | 5.5 (16) | 4.3 (9)

4. Secondary Outcome: Range of Knee Flexion
Description: Range of knee flexion for active motion will be recorded at 3 week follow-up for all groups. The greater range of motion the better, with a good outcome considered at least 115 degrees of motion.
Time Frame: Postoperative day 21
Measure: Mean (Standard Deviation); unit: degrees
Groups:
- Adductor Canal Block: 15 cc's of 0.5% bupivacaine preoperatively administered by the regional pain anesthesia team in the pre-operative block area, just prior to surgery.
  Adductor Canal Block (ACB)
  Bupivacaine: 15 cc's of 0.5% bupivacaine or 50 cc's short-acting bupivacaine (SB), intramuscular injection
Arm/Group | Adductor Canal Block | Periarticular SB | ACB + SB
Number analyzed (Participants) | 53 | 51 | 51
degrees | 99 (15) | 104 (12) | 101 (16)

5. Secondary Outcome: Length of Hospital Stay
Description: Total length of hospital stay from time of surgery through time of discharge will be recorded. The shorter the length of stay (days) the better. Range 0 days to 5 days.
Time Frame: Up to Day 5
Measure: Mean (Standard Deviation); unit: days
Groups:
- ACB + SB: 15 cc's of 0.5% bupivacaine preoperatively administered by the regional pain anesthesia team in the pre-operative block area, just prior to surgery.
  50 cc's of bupivacaine will be injected intraoperatively, just prior to wound closure, by the performing surgeon.
  Bupivacaine: 15 cc's of 0.5% bupivacaine or50 cc's short-acting bupivacaine (SB), intramuscular injection
Arm/Group | Adductor Canal Block | Periarticular SB | ACB + SB
Number analyzed (Participants) | 53 | 51 | 51
days | 2.9 (1.5) | 2.5 (1.2) | 2.5 (2.1)

ADVERSE EVENTS:
Time Frame: postoperative day 0 through post-operative day 21.
Description: No serious adverse events, including mortality. This was a healthy cohort of patients undergoing elective surgery for total knee replacement. There were no expected adverse events.
Groups:
- Adductor Canal Block: 15 cc's of 0.5% bupivacaine preoperatively administered by the regional pain anesthesia team in the pre-operative block area, just prior to surgery.
  Adductor Canal Block (ACB)
  Bupivacaine: 15 cc's of 0.5% bupivacaine or 50 cc's of 0.25% short-acting bupivacaine (SB), intramuscular injection
- ACB + SB: 15 cc's of 0.5% bupivacaine preoperatively administered by the regional pain anesthesia team in the pre-operative block area, just prior to surgery.
  50 cc's of 0.25% bupivacaine will be injected intraoperatively, just prior to wound closure, by the performing surgeon.
  Bupivacaine: 15 cc's of 0.5% bupivacaine or 50 cc's of 0.25% short-acting bupivacaine (SB), intramuscular injection
Arm/Group | Adductor Canal Block | Periarticular SB | ACB + SB
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/51 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/51 | 0/51
Other Adverse Events (participants affected / at risk) | 0/53 | 0/51 | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-01): https://cdn.clinicaltrials.gov/large-docs/49/NCT02777749/Prot_SAP_000.pdf